CLINICAL TRIAL: NCT01604109
Title: Effect of CPP-ACP Paste on Dental Caries in Primary Teeth: A Randomized Trial
Brief Title: Effect of CPP-ACP Paste on Dental Caries in Primary Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Thanya Sitthisettapong, Faculty of Dentistry, Thammasat University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TU-Dent-01; D43TW007768 (NIH)
Record Dates: First submitted 2012-05-19; First posted 2012-05-23 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-06

CONDITIONS: Dental Caries
Keywords: Caries detection/diagnosis/prevention; Preventive Dentistry; Casien Phosphopeptide; Remineralization; Clinical trial
MeSH Terms: conditions — Dental Caries | interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tooth Mousse (Active Comparator): 10% w/v Calcium Phosphopeptide Amorphous Calcium Phosphate paste
  Interventions: Drug: 10 % w/v CPP-ACP paste
- placebo control paste (Placebo Comparator): the paste without Calcium phosphopeptide - Amorphous Calcium Phosphate
  Interventions: Drug: the paste without CPP-ACP

INTERVENTIONS:
Drug: 10 % w/v CPP-ACP paste — Apply once a day at school by school teacher, following fluoride toothbrushing after lunch
  Other Names: Tooth Mousse
  Arms: Tooth Mousse
Drug: the paste without CPP-ACP — Apply once a day at school by school teacher, following fluoride toothbrushing after lunch.
  Arms: placebo control paste

SUMMARY:
The purpose of this study is to determine if adding daily application of CPP-ACP containing paste for one year is superior to regular fluoride tooth brushing in preventing dental caries in high caries risk Thai preschool children.

DETAILED DESCRIPTION:
The 6th National Oral Health Survey in Thailand 2006-2007 reported that 3-year-old children who resided in central part have the highest dental caries prevalence of 69.8 percent with dmft affecting 3.63 teeth on average. Fluoride is widely accepted as the most effective tool to caries prevention for initial caries lesions. Current best practice recommends twice-daily tooth brushing with fluoride toothpaste for dentate children.

CPP-ACP can bolster the effects of fluoridated toothpaste alone to prevent caries.Currently, almost all clinical trials have investigated the effectiveness of CPP-ACP containing products in dental caries prevention and enhancing remineralization of initial carious lesion in the permanent dentition of young adolescents. There are no clinical studies of the effect of a CPP-ACP containing product to prevent dental caries in the primary dentition of young children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Thai boys and girl aged between 2 1/2 - 3 1/2
* Normal development of dentition
* Diagnosed as high caries risk by using the Caries-risk Assessment Tool(CAT)

Exclusion Criteria:

* Chronic use of medications or antibiotics.
* Lack of cooperation in oral examination
* Milk protein allergy and/or benzoate preservatives
* Presence at baseline oral soft tissue lesion and enamel hypoplasia.
* Receive fluoride supplement and professional topical fluoride application at least three months before the beginning of study or during study period

Ages: 30 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 296 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanya Sitthisettapong, Principal Investigator — Faculty of Dentistry, Thammasat University
Locations (1):
- Faculty of Dentistry, Thammasat University, Klongluang, Patumthani, Thailand

REFERENCES:
- [Derived] Sitthisettapong T, Phantumvanit P, Huebner C, Derouen T. Effect of CPP-ACP paste on dental caries in primary teeth: a randomized trial. J Dent Res. 2012 Sep;91(9):847-52. doi: 10.1177/0022034512454296. Epub 2012 Jul 17. PMID 22805294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place in the central part of Thailand, where water [F]<0.1 ppm. The recruitment began in June 2010. There were 304 healthy Thai boys and girls from ten public nursery schools enrolled in the study. The baseline examination was performed at school in July-August, 2010.
Pre-assignment Details: Six children were excluded from the study because they did not complete the inclusion criteria: autism (1), milk protein allergy (1), taking fluoride table (1), and no high caries risk (3).
Groups:
- Tooth Mousse: 10% w/v Calcium Phosphopeptide Amorphous Calcium Phosphate paste
  10 % w/v CPP-ACP paste : Apply once a day at school by school teacher, following fluoride toothbrushing after lunch
- Placebo Control Paste: the paste without Calcium phosphopeptide - Amorphous Calcium Phosphate
  the paste without CPP-ACP : Apply once a day at school by school teacher, following fluoride toothbrushing after lunch.
Period: Overall Study
Arm/Group | Tooth Mousse | Placebo Control Paste
Started | 150 | 146
Completed | 117 | 112
Not Completed | 33 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tooth Mousse | Placebo Control Paste | Total
Number analyzed (Participants) | 150 | 146 | 296
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 150 | 146 | 296
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3.08 (0.24) | 3.10 (0.25) | 3.09 (0.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 153
  Male | 72 | 71 | 143
Region of Enrollment [Number; unit: participants]
  Thailand | 150 | 146 | 296

OUTCOME MEASURES:

1. Primary Outcome: the Mean Number of Enamel Carious Lesion
Description: tooth surface that was classified as ICDAS code 1-3
Time Frame: one calender year
Measure: Mean (Standard Deviation); unit: Surfaces
Arm/Group | Tooth Mousse | Placebo Control Paste
Number analyzed (Participants) | 150 | 146
Surfaces | 13.69 (7.94) | 14.55 (9.56)

2. Secondary Outcome: Quantitative Light-induced Fluorescence (QLF) Parameters
Description: percent fluorescence loss, lesion area, lesion volume
Time Frame: one calender year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Tooth Mousse | Placebo Control Paste
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/146
Other Adverse Events (participants affected / at risk) | 0/150 | 0/146

LIMITATIONS AND CAVEATS:
This one year study was performed on high caries risk pre-school children who enrolled in government nursery schools in central part of Thailand.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No